CLINICAL TRIAL: NCT05016505
Title: A Randomized Controlled Trial to Support Smoke-Free Policy Compliance in Public Housing
Brief Title: Supporting Smoke-Free Policy Compliance in Public Housing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Diana Hernandez, PhD, Associate Professor of Sociomedical Sciences, Columbia University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: AAAT1493; R01CA240555-01A1 (NIH)
Record Dates: First submitted 2021-07-20; First posted 2021-08-23 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Smoking; Smoking Cessation; Smoking Reduction; Smoking Behaviors
Keywords: smoking; secondhand smoke
MeSH Terms: conditions — Smoking; Smoking Cessation; Smoking Reduction

STUDY DESIGN:
Intervention Model Description: The proposed design will be a borough-stratified, four-arm, factorial-design, cluster RCT that will target 64 randomly selected buildings (16 buildings per arm) in separate New York City Housing Authority (NYCHA) developments.
  The investigators will recruit and follow 8 randomly selected residents stratified by smoking status- 4 smokers and 4 non-smokers- per building (n=512 residents) into four arms: (1) reduction (relocation and reduction in personal smoking)/cessation, (2) resident endorsement, (3) reduction (relocation and reduction in personal smoking)/cessation plus resident endorsement and (4) the standard approach (128 participants per arm).
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Compliance through reduction (relocation and reduction of personal smoking) and cessation (Experimental): Smokers will be referred by the survey team to peer educators from a community-based organization trained to provide peer to peer health education including tobacco cessation support. The peer educator will coordinate smoking cessation support, including serving as a liaison between participant and research team, providing information regarding the smoke-free policy and opportunities for relocation, and connecting participant to access to tobacco replacement therapy and/or physician support if deemed appropriate.
  Interventions: Behavioral: Reduction (relocation and reduction of personal smoking) and cessation
- Compliance through resident endorsement (Experimental): Buildings assigned will be targeted for a series of 2 in-residence programs that involve community forums and the creative arts to garner resident endorsements of smoke-free living environments. Premised on resident engagement, this arm seeks to impact social and physical dimensions of the residential environment to achieve compliance. The sessions will: 1) inform residents of risks associated with smoking and secondhand smoke; 2) identify reasons to have a smoke-free home, 3) ask residents to sign a pledge on paper and/or virtually; 4) display smoke-free signage on doors and/or social media pages with an original hashtag (#Smokefree[building address]); and 5) refer residents to the Smoke-free NYCHA website for information on the policy and existing cessation resources.
  Interventions: Behavioral: Resident Endorsement
- Compliance through reduction/cessation plus resident endorsement (combined) (Experimental): The combined intervention will be carried out in the buildings assigned to this RCT arm, which will provide in-residence programs based on the resident endorsement treatment and the smoking relocation/cessation treatment. Both will occur simultaneously with one geared toward all building residents (resident endorsement) and the other targeting smokers (smoking relocation/cessation) with the goal of reducing both personal smoking and secondhand smoke exposure.
  Interventions: Behavioral: Reduction (relocation and reduction of personal smoking) and cessation; Behavioral: Resident Endorsement
- Standard NYCHA approach (control) (No Intervention): Buildings and study participants assigned to this arm will be recruited and followed over a 12-month period to assess outcomes. No additional programs or services will be delivered to the buildings or residents assigned to this arm beyond standard programs that NYCHA may provide to support the smoke-free mandate. Field staff will document any policy-related signage, activities or information to which these participants are exposed.

INTERVENTIONS:
Behavioral: Reduction (relocation and reduction of personal smoking) and cessation — Individual-level. Peer educator to provide reduction/cessation and/or relocation support.
  Arms: Compliance through reduction (relocation and reduction of personal smoking) and cessation; Compliance through reduction/cessation plus resident endorsement (combined)
Behavioral: Resident Endorsement — Building-level. Peer educator to conduct building-level sessions.
  Arms: Compliance through reduction/cessation plus resident endorsement (combined); Compliance through resident endorsement

SUMMARY:
This project seeks to determine the effectiveness of two types of interventions to reduce exposure to secondhand smoke in residential buildings. One intervention is geared toward all building residents (resident endorsement) and the other targets smokers (smoking reduction via relocation and reduction in personal smoking/cessation) with the goal of reducing personal smoking and secondhand smoke exposure.

DETAILED DESCRIPTION:
Smoke-free housing policies in multi-unit housing are promising and increasingly widespread interventions to reduce smoking and secondhand smoke exposure. Little research has identified factors that improve compliance with smoke-free housing policies in low-income multi-unit housing and test corresponding solutions.

The proposed randomized controlled trial (RCT) addresses key gaps in knowledge and capitalizes on key scientific opportunities by: 1) leveraging the federal mandate to ban smoking in a public housing system of more than sufficient size to conduct an adequately powered RCT; 2) expanding our understanding of smoke-free policy compliance beyond policy implementation by testing two novel treatments: a) in-residence smoking cessation and b) resident endorsement, while 3) addressing population and location-specific tobacco-related disparities.

The investigators hypothesize that the relocation/cessation plus resident endorsement intervention will yield significantly larger reductions in personal smoking and secondhand smoke exposure, compared to standalone interventions and the standard approach.

ELIGIBILITY:
Building Inclusion Criteria:

* NYCHA buildings in Manhattan & the Bronx (stratified evenly by borough) with more than 50 units, not undergoing major renovations.

Building Exclusion Criteria:

* Buildings in a borough that is not in Manhattan or the Bronx
* Buildings smaller than 50 units
* Buildings undergoing major renovations
* Buildings that are or will be part of Rental Assistance Demonstration (RAD) or Permanent Affordability Commitment Together (PACT)
* Buildings that are mixed finance
* Buildings that are exclusively for elderly
* Buildings that are privately managed
* Buildings that have other research studies ongoing

Participant Inclusion Criteria:

* Recruit NYCHA residents via door knocking and lobby intercepts until we reach our targeted number per group (4 smokers, 4 non-smokers in each building).
* Residents will be screened for smoking status. Both smokers and non-smokers to be recruited but only one participant- smoker or a non-smoker- will be recruited per apartment.
* Smoking will be defined as those that report using a cigarette or other combustible tobacco product (e.g., little cigar, cigarillo) at least 5 days in the past month. Non-smokers include never smokers and former smokers who had quit 12 months ago or earlier.
* Additional eligibility criteria include individuals above 18 years old living in the building at least 5 days/week and 9 months/year, not planning on moving in the next 2 years.

Participant Exclusion Criteria:

* Individuals with severe physical or mental medical conditions (i.e. cognitive disability) or other factors that could limit participation or ability to give informed consent in the study at baseline or during follow-ups.
* Individuals who participated in the earlier focus groups.
* Individuals who only smoke non-tobacco products (e.g., marijuana).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 405 (Actual)
Dates: Start 2022-02-03 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Change in number of cigarettes smoked per day | Measured at baseline (in person interview), 3 months (phone interview) and 12 months (in person interview)
  Self-reported average number of cigarettes smoked per day among smokers
Change in salivary cotinine | At baseline and at the 12-month follow-up
  Salivary cotinine (saliva collected as passive drool) will be measured for 25% of the sample among smokers and non-smokers alike
Change in secondhand smoke exposure | Measured at baseline (in person interview), 3 months (phone interview) and 12 months (in person interview)
  Self-reported secondhand smoking exposure (hours of secondhand smoke exposure in the building in the past 7 days); among smokers & non-smokers

SECONDARY OUTCOMES:
Change in number of participants with successful quit attempts | Measured at baseline (in person interview), 3 months (phone interview) and 12 months (in person interview)
  Binary; whether smokers have successfully quit
Change in number of quit attempts | Measured at baseline (in person interview), 3 months (phone interview) and 12 months (in person interview)
  Mean number of quitting attempts among smokers
Change in number of participants with secondhand smoke observations | Ever observing someone smoking indoors within the past 7 days measured at baseline (in person interview), 3 months (phone interview) and 12 months (in person interview)
  Binary; whether participant has observed someone smoking indoors in the building; among smokers & non-smokers
Change in number of hours of secondhand smoke exposure | Number of hours observed someone smoking indoors within the past 7 days measured at baseline (in person interview), 3 months (phone interview) and 12 months (in person interview)
  Counted number of hours of exposure
Change in number of smokers | At each building visit at baseline and 12 months
  Counted number of people observed smoking in common areas
Change in number of cigarette butts | At each building visit at baseline and 12 months
  Counted number of cigarette butts observed in common areas

CONTACTS AND LOCATIONS:
Overall Officials: Diana Hernández, PhD, Principal Investigator — Associate Professor of Sociomedical Sciences
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Data from approximately 512 participants will be released to sponsor (NIH) once the final dataset is analyzed and main findings are accepted for publication to support and validate study findings. This will include participant demographics, data from interviews, and laboratory data from saliva samples. Identifiers might be removed from the identifiable private information or identifiable biospecimens and that, after such removal, the information or biospecimens could be used for future research studies without additional consent from the subject. De-identified participant data may be utilized for the purposes of repeated analyses by other researchers to verify findings, and/or to promote further research with new or alternative hypotheses. The mechanism of distribution will be a data sharing agreement.
Time Frame: Data will be available once the final dataset is analyzed and main findings are accepted for publication to support and validate study findings.
  Access will be granted for researchers, institutions, and/or the broader public for as long as the data is anticipated to be useful. With the data sharing agreement in mind, the data can be made available for the duration of time needed to conduct analyses.
Access Criteria: Access should be granted to those with a reputable background in the scientific field who have either a scientific or medical degree and/or a relevant position to ask for the data. Individuals should also express their intended use of the data. These requests will be routinely reviewed by the principal investigator [and/or designated team member].

REFERENCES:
- [Background] Branas CC, Culhane D, Richmond TS, Wiebe DJ. Novel Linkage of Individual and Geographic Data to Study Firearm Violence. Homicide Stud. 2008 Aug;12(3):298-320. doi: 10.1177/1088767908319756. PMID 20617158
- [Background] Kim S, Apelberg BJ, Avila-Tang E, Hepp L, Yun D, Samet JM, Breysse PN. Utility and cutoff value of hair nicotine as a biomarker of long-term tobacco smoke exposure, compared to salivary cotinine. Int J Environ Res Public Health. 2014 Aug 15;11(8):8368-82. doi: 10.3390/ijerph110808368. PMID 25153466
- [Background] Sims M, Mindell JS, Jarvis MJ, Feyerabend C, Wardle H, Gilmore A. Did smokefree legislation in England reduce exposure to secondhand smoke among nonsmoking adults? Cotinine analysis from the Health Survey for England. Environ Health Perspect. 2012 Mar;120(3):425-30. doi: 10.1289/ehp.1103680. Epub 2011 Dec 12. PMID 22169225
- [Background] Kondo MC, Bream KD, Barg FK, Branas CC. A random spatial sampling method in a rural developing nation. BMC Public Health. 2014 Apr 10;14:338. doi: 10.1186/1471-2458-14-338. PMID 24716473
- [Background] Wong MS, Grande DT, Mitra N, Radhakrishnan A, Branas CC, Ward KR, Pollack CE. Racial Differences in Geographic Access to Medical Care as Measured by Patient Report and Geographic Information Systems. Med Care. 2017 Sep;55(9):817-822. doi: 10.1097/MLR.0000000000000774. PMID 28731892
- [Background] Winickoff JP, Gottlieb M, Mello MM. Regulation of smoking in public housing. N Engl J Med. 2010 Jun 17;362(24):2319-25. doi: 10.1056/NEJMhle1000941. No abstract available. PMID 20554988
- [Background] King BA, Travers MJ, Cummings KM, Mahoney MC, Hyland AJ. Secondhand smoke transfer in multiunit housing. Nicotine Tob Res. 2010 Nov;12(11):1133-41. doi: 10.1093/ntr/ntq162. Epub 2010 Oct 1. PMID 20889473
- [Background] Kraev TA, Adamkiewicz G, Hammond SK, Spengler JD. Indoor concentrations of nicotine in low-income, multi-unit housing: associations with smoking behaviours and housing characteristics. Tob Control. 2009 Dec;18(6):438-44. doi: 10.1136/tc.2009.029728. Epub 2009 Aug 13. PMID 19679890
- [Background] King BA, Babb SD, Tynan MA, Gerzoff RB. National and state estimates of secondhand smoke infiltration among U.S. multiunit housing residents. Nicotine Tob Res. 2013 Jul;15(7):1316-21. doi: 10.1093/ntr/nts254. Epub 2012 Dec 17. PMID 23248030
- [Background] Office on Smoking and Health (US). The Health Consequences of Involuntary Exposure to Tobacco Smoke: A Report of the Surgeon General. Atlanta (GA): Centers for Disease Control and Prevention (US); 2006. Available from http://www.ncbi.nlm.nih.gov/books/NBK44324/ PMID 20669524
- [Background] Nguyen KH, Gomez Y, Homa DM, King BA. Tobacco Use, Secondhand Smoke, and Smoke-Free Home Rules in Multiunit Housing. Am J Prev Med. 2016 Nov;51(5):682-692. doi: 10.1016/j.amepre.2016.05.009. Epub 2016 Jul 13. PMID 27423656
- [Background] Snyder K, Vick JH, King BA. Smoke-free multiunit housing: a review of the scientific literature. Tob Control. 2016 Jan;25(1):9-20. doi: 10.1136/tobaccocontrol-2014-051849. Epub 2015 Jan 7. PMID 25566811
- [Background] Jamal A, Agaku IT, O'Connor E, King BA, Kenemer JB, Neff L. Current cigarette smoking among adults--United States, 2005-2013. MMWR Morb Mortal Wkly Rep. 2014 Nov 28;63(47):1108-12. PMID 25426653
- [Background] Helms VE, King BA, Ashley PJ. Cigarette smoking and adverse health outcomes among adults receiving federal housing assistance. Prev Med. 2017 Jun;99:171-177. doi: 10.1016/j.ypmed.2017.02.001. Epub 2017 Feb 10. PMID 28192095
- [Background] Brown N, Luckett T, Davidson PM, Di Giacomo M. Interventions to reduce harm from smoking with families in infancy and early childhood: a systematic review. Int J Environ Res Public Health. 2015 Mar 16;12(3):3091-119. doi: 10.3390/ijerph120303091. PMID 25785496
- [Background] Homa DM, Neff LJ, King BA, Caraballo RS, Bunnell RE, Babb SD, Garrett BE, Sosnoff CS, Wang L; Centers for Disease Control and Prevention (CDC). Vital signs: disparities in nonsmokers' exposure to secondhand smoke--United States, 1999-2012. MMWR Morb Mortal Wkly Rep. 2015 Feb 6;64(4):103-8. PMID 25654612
- [Background] Stapleton M, Howard-Thompson A, George C, Hoover RM, Self TH. Smoking and asthma. J Am Board Fam Med. 2011 May-Jun;24(3):313-22. doi: 10.3122/jabfm.2011.03.100180. PMID 21551404
- [Background] Stein A, Suttie J, Baker L, Agans R, Xue W, Bowling JM. Predictors of smoke-free policies in affordable multiunit housing, North Carolina, 2013. Prev Chronic Dis. 2015 May 14;12:E73. doi: 10.5888/pcd12.140506. PMID 25974143
- [Background] Lee JG, Henriksen L, Rose SW, Moreland-Russell S, Ribisl KM. A Systematic Review of Neighborhood Disparities in Point-of-Sale Tobacco Marketing. Am J Public Health. 2015 Sep;105(9):e8-18. doi: 10.2105/AJPH.2015.302777. Epub 2015 Jul 16. PMID 26180986
- [Background] Ribisl KM, D'Angelo H, Feld AL, Schleicher NC, Golden SD, Luke DA, Henriksen L. Disparities in tobacco marketing and product availability at the point of sale: Results of a national study. Prev Med. 2017 Dec;105:381-388. doi: 10.1016/j.ypmed.2017.04.010. Epub 2017 Apr 6. PMID 28392252
- [Background] Feinberg A, Lopez PM, Wyka K, Islam N, Seidl L, Drackett E, Mata A, Pinzon J, Baker MR, Lopez J, Trinh-Shevrin C, Shelley D, Bailey Z, Maybank KA, Thorpe LE. Prevalence and Correlates of Smoking among Low-Income Adults Residing in New York City Public Housing Developments-2015. J Urban Health. 2017 Aug;94(4):525-533. doi: 10.1007/s11524-017-0180-z. PMID 28656541
- [Background] Farley SM, Schroth KR, Curtis CJ, Angell S. Evidence of Support for Smoke-Free Public Housing Among New York City Residents. Public Health Rep. 2016 Jan-Feb;131(1):2-3. doi: 10.1177/003335491613100102. No abstract available. PMID 26843660
- [Background] Rogers ES, Vargas EA. Tobacco retail environment near housing programmes for patients with mental health conditions in New York City. Tob Control. 2018 Sep;27(5):526-533. doi: 10.1136/tobaccocontrol-2016-053590. Epub 2017 Aug 30. PMID 28855299
- [Background] Parton HB, Greene R, Flatley AM, Viswanathan N, Wilensky L, Berman J, Schneider AE, Uribe A, Olson EC, Waddell EN, Thorpe LE. Health of older adults in New York City public housing: part 1, findings from the New York City Housing Authority Senior Survey. Care Manag J. 2012;13(3):134-47. doi: 10.1891/1521-0987.13.3.134. No abstract available. PMID 23072177
- [Background] Albers AB, Siegel M, Cheng DM, Biener L, Rigotti NA. Relation between local restaurant smoking regulations and attitudes towards the prevalence and social acceptability of smoking: a study of youths and adults who eat out predominantly at restaurants in their town. Tob Control. 2004 Dec;13(4):347-55. doi: 10.1136/tc.2003.007336. PMID 15564617
- [Background] Haw SJ, Gruer L. Changes in exposure of adult non-smokers to secondhand smoke after implementation of smoke-free legislation in Scotland: national cross sectional survey. BMJ. 2007 Sep 15;335(7619):549. doi: 10.1136/bmj.39315.670208.47. Epub 2007 Sep 9. PMID 17827485
- [Background] Hopkins DP, Razi S, Leeks KD, Priya Kalra G, Chattopadhyay SK, Soler RE; Task Force on Community Preventive Services. Smokefree policies to reduce tobacco use. A systematic review. Am J Prev Med. 2010 Feb;38(2 Suppl):S275-89. doi: 10.1016/j.amepre.2009.10.029. PMID 20117612
- [Background] Cheng KW, Glantz SA, Lightwood JM. Association between smokefree laws and voluntary smokefree-home rules. Am J Prev Med. 2011 Dec;41(6):566-72. doi: 10.1016/j.amepre.2011.08.014. PMID 22099232
- [Background] Hahn EJ. Smokefree legislation: a review of health and economic outcomes research. Am J Prev Med. 2010 Dec;39(6 Suppl 1):S66-76. doi: 10.1016/j.amepre.2010.08.013. PMID 21074680
- [Background] Klepeis NE, Nelson WC, Ott WR, Robinson JP, Tsang AM, Switzer P, Behar JV, Hern SC, Engelmann WH. The National Human Activity Pattern Survey (NHAPS): a resource for assessing exposure to environmental pollutants. J Expo Anal Environ Epidemiol. 2001 May-Jun;11(3):231-52. doi: 10.1038/sj.jea.7500165. PMID 11477521
- [Background] Bohac DL, Hewett MJ, Hammond SK, Grimsrud DT. Secondhand smoke transfer and reductions by air sealing and ventilation in multiunit buildings: PFT and nicotine verification. Indoor Air. 2011 Feb;21(1):36-44. doi: 10.1111/j.1600-0668.2010.00680.x. PMID 20846212
- [Background] National Center for Chronic Disease Prevention and Health Promotion (US) Office on Smoking and Health. The Health Consequences of Smoking-50 Years of Progress: A Report of the Surgeon General. Atlanta (GA): Centers for Disease Control and Prevention (US); 2014. Available from http://www.ncbi.nlm.nih.gov/books/NBK179276/ PMID 24455788
- [Background] Chambers C, Sung HY, Max W. Home exposure to secondhand smoke among people living in multiunit housing and single family housing: a study of California adults, 2003-2012. J Urban Health. 2015 Apr;92(2):279-90. doi: 10.1007/s11524-014-9919-y. PMID 25466438
- [Background] Kennedy RD, Ellens-Clark S, Nagge L, Douglas O, Madill C, Kaufman P. A Smoke-Free Community Housing Policy: Changes in Reported Smoking Behaviour-Findings from Waterloo Region, Canada. J Community Health. 2015 Dec;40(6):1207-15. doi: 10.1007/s10900-015-0050-0. PMID 26070870
- [Background] Kingsbury JH, Reckinger D. Clearing the Air: Smoke-Free Housing Policies, Smoking, and Secondhand Smoke Exposure Among Affordable Housing Residents in Minnesota, 2014-2015. Prev Chronic Dis. 2016 Aug 18;13:E111. doi: 10.5888/pcd13.160195. PMID 27536903
- [Background] Pizacani BA, Maher JE, Rohde K, Drach L, Stark MJ. Implementation of a smoke-free policy in subsidized multiunit housing: effects on smoking cessation and secondhand smoke exposure. Nicotine Tob Res. 2012 Sep;14(9):1027-34. doi: 10.1093/ntr/ntr334. Epub 2012 Feb 7. PMID 22318686
- [Background] Young W, Karp S, Bialick P, Liverance C, Seder A, Berg E, Karp L. Health, Secondhand Smoke Exposure, and Smoking Behavior Impacts of No-Smoking Policies in Public Housing, Colorado, 2014-2015. Prev Chronic Dis. 2016 Oct 20;13:E148. doi: 10.5888/pcd13.160008. PMID 27763830
- [Background] Russo ET, Hulse TE, Adamkiewicz G, Levy DE, Bethune L, Kane J, Reid M, Shah SN. Comparison of indoor air quality in smoke-permitted and smoke-free multiunit housing: findings from the Boston Housing Authority. Nicotine Tob Res. 2015 Mar;17(3):316-22. doi: 10.1093/ntr/ntu146. Epub 2014 Aug 25. PMID 25156526
- [Background] Jackson SL, Bonnie RJ. A systematic examination of smoke-free policies in multiunit dwellings in Virginia as reported by property managers: implications for prevention. Am J Health Promot. 2011 Sep-Oct;26(1):37-44. doi: 10.4278/ajhp.091005-QUAN-329. PMID 21879941
- [Background] Baezconde-Garbanati LA, Weich-Reushe K, Espinoza L, Portugal C, Barahona R, Garbanati J, Seedat F, Unger JB. Secondhand smoke exposure among Hispanics/Latinos living in multiunit housing: exploring barriers to new policies. Am J Health Promot. 2011 May-Jun;25(5 Suppl):S82-90. doi: 10.4278/ajhp.100628-QUAL-219. PMID 21510793
- [Background] Ballor DL, Henson H, MacGuire K. Support for no-smoking policies among residents of public multiunit housing differs by smoking status. J Community Health. 2013 Dec;38(6):1074-80. doi: 10.1007/s10900-013-9716-7. PMID 23775035
- [Background] Hennrikus D, Pentel PR, Sandell SD. Preferences and practices among renters regarding smoking restrictions in apartment buildings. Tob Control. 2003 Jun;12(2):189-94. doi: 10.1136/tc.12.2.189. PMID 12773730
- [Background] Hewett MJ, Sandell SD, Anderson J, Niebuhr M. Secondhand smoke in apartment buildings: renter and owner or manager perspectives. Nicotine Tob Res. 2007 Jan;9 Suppl 1:S39-47. doi: 10.1080/14622200601083442. PMID 17365725
- [Background] Hewett MJ, Ortland WH, Brock BE, Heim CJ. Secondhand smoke and smokefree policies in owner-occupied multi-unit housing. Am J Prev Med. 2012 Nov;43(5 Suppl 3):S187-96. doi: 10.1016/j.amepre.2012.07.039. PMID 23079216
- [Background] Hood NE, Ferketich AK, Klein EG, Wewers ME, Pirie P. Individual, social, and environmental factors associated with support for smoke-free housing policies among subsidized multiunit housing tenants. Nicotine Tob Res. 2013 Jun;15(6):1075-83. doi: 10.1093/ntr/nts246. Epub 2012 Nov 7. PMID 23136269
- [Background] Lortet-Tieulent J, Goding Sauer A, Siegel RL, Miller KD, Islami F, Fedewa SA, Jacobs EJ, Jemal A. State-Level Cancer Mortality Attributable to Cigarette Smoking in the United States. JAMA Intern Med. 2016 Dec 1;176(12):1792-1798. doi: 10.1001/jamainternmed.2016.6530. PMID 27775761
- [Background] Jamal A, King BA, Neff LJ, Whitmill J, Babb SD, Graffunder CM. Current Cigarette Smoking Among Adults - United States, 2005-2015. MMWR Morb Mortal Wkly Rep. 2016 Nov 11;65(44):1205-1211. doi: 10.15585/mmwr.mm6544a2. PMID 27832052
- [Background] King BA, Hyland AJ, Borland R, McNeill A, Cummings KM. Socioeconomic variation in the prevalence, introduction, retention, and removal of smoke-free policies among smokers: findings from the International Tobacco Control (ITC) Four Country Survey. Int J Environ Res Public Health. 2011 Feb;8(2):411-34. doi: 10.3390/ijerph8020411. Epub 2011 Jan 31. PMID 21556194
- [Background] Clegg LX, Reichman ME, Miller BA, Hankey BF, Singh GK, Lin YD, Goodman MT, Lynch CF, Schwartz SM, Chen VW, Bernstein L, Gomez SL, Graff JJ, Lin CC, Johnson NJ, Edwards BK. Impact of socioeconomic status on cancer incidence and stage at diagnosis: selected findings from the surveillance, epidemiology, and end results: National Longitudinal Mortality Study. Cancer Causes Control. 2009 May;20(4):417-35. doi: 10.1007/s10552-008-9256-0. Epub 2008 Nov 12. PMID 19002764
- [Background] Siegel R, Ward E, Brawley O, Jemal A. Cancer statistics, 2011: the impact of eliminating socioeconomic and racial disparities on premature cancer deaths. CA Cancer J Clin. 2011 Jul-Aug;61(4):212-36. doi: 10.3322/caac.20121. Epub 2011 Jun 17. PMID 21685461
- [Background] Steenland K, Henley J, Thun M. All-cause and cause-specific death rates by educational status for two million people in two American Cancer Society cohorts, 1959-1996. Am J Epidemiol. 2002 Jul 1;156(1):11-21. doi: 10.1093/aje/kwf001. PMID 12076884
- [Background] Tobacco use among U.S. racial/ethnic minority groups--African Americans, American Indians and Alaska Natives, Asian Americans and Pacific Islanders, Hispanics. A Report of the Surgeon General. Executive summary. MMWR Recomm Rep. 1998 Oct 9;47(RR-18):v-xv, 1-16. No abstract available. PMID 9784089
- [Background] Branas CC, Macdonald JM. A simple strategy to transform health, all over the place. J Public Health Manag Pract. 2014 Mar-Apr;20(2):157-9. doi: 10.1097/PHH.0000000000000051. No abstract available. PMID 24458312
- [Background] Bauer UE, Briss PA, Goodman RA, Bowman BA. Prevention of chronic disease in the 21st century: elimination of the leading preventable causes of premature death and disability in the USA. Lancet. 2014 Jul 5;384(9937):45-52. doi: 10.1016/S0140-6736(14)60648-6. Epub 2014 Jul 1. PMID 24996589
- [Background] Yen IH, Syme SL. The social environment and health: a discussion of the epidemiologic literature. Annu Rev Public Health. 1999;20:287-308. doi: 10.1146/annurev.publhealth.20.1.287. PMID 10352860
- [Background] Schroeder SA. Shattuck Lecture. We can do better--improving the health of the American people. N Engl J Med. 2007 Sep 20;357(12):1221-8. doi: 10.1056/NEJMsa073350. No abstract available. PMID 17881753
- [Background] Centers for Disease Control and Prevention (CDC). Ten great public health achievements--United States, 1900-1999. MMWR Morb Mortal Wkly Rep. 1999 Apr 2;48(12):241-3. PMID 10220250
- [Background] Committee on Valuing Community-Based, Non-Clinical Prevention Programs; Board on Population Health and Public Health Practice; Institute of Medicine. An Integrated Framework for Assessing the Value of Community-Based Prevention. Washington (DC): National Academies Press (US); 2012 Oct 29. Available from http://www.ncbi.nlm.nih.gov/books/NBK206926/ PMID 24901190
- [Background] Garrett BE, Dube SR, Babb S, McAfee T. Addressing the Social Determinants of Health to Reduce Tobacco-Related Disparities. Nicotine Tob Res. 2015 Aug;17(8):892-7. doi: 10.1093/ntr/ntu266. Epub 2014 Dec 16. PMID 25516538
- [Background] Cokkinides V, Bandi P, McMahon C, Jemal A, Glynn T, Ward E. Tobacco control in the United States--recent progress and opportunities. CA Cancer J Clin. 2009 Nov-Dec;59(6):352-65. doi: 10.3322/caac.20037. PMID 19897839
- [Background] Barnoya J, Glantz S. Association of the California tobacco control program with declines in lung cancer incidence. Cancer Causes Control. 2004 Sep;15(7):689-95. doi: 10.1023/B:CACO.0000036187.13805.30. PMID 15280627
- [Background] Chaloupka FJ, Pacula RL. Sex and race differences in young people's responsiveness to price and tobacco control policies. Tob Control. 1999 Winter;8(4):373-7. doi: 10.1136/tc.8.4.373. PMID 10629242
- [Background] Baker SP. Childhood injuries: the community approach to prevention. J Public Health Policy. 1981 Sep;2(3):235-46. No abstract available. PMID 7298840
- [Background] Frieden TR. A framework for public health action: the health impact pyramid. Am J Public Health. 2010 Apr;100(4):590-5. doi: 10.2105/AJPH.2009.185652. Epub 2010 Feb 18. PMID 20167880
- [Background] Rise J, Kovac V, Kraft P, Moan IS. Predicting the intention to quit smoking and quitting behaviour: extending the theory of planned behaviour. Br J Health Psychol. 2008 May;13(Pt 2):291-310. doi: 10.1348/135910707X187245. Epub 2007 Mar 5. PMID 17535498
- [Background] Norman P, Conner M, Bell R. The theory of planned behavior and smoking cessation. Health Psychol. 1999 Jan;18(1):89-94. doi: 10.1037//0278-6133.18.1.89. PMID 9925050
- [Background] Godin G, Kok G. The theory of planned behavior: a review of its applications to health-related behaviors. Am J Health Promot. 1996 Nov-Dec;11(2):87-98. doi: 10.4278/0890-1171-11.2.87. PMID 10163601
- [Background] Macy JT, Middlestadt SE, Seo DC, Kolbe LJ, Jay SJ. Applying the theory of planned behavior to explore the relation between smoke-free air laws and quitting intentions. Health Educ Behav. 2012 Feb;39(1):27-34. doi: 10.1177/1090198111404702. Epub 2011 Apr 25. PMID 21518919
- [Background] Giordano GN, Lindstrom M. The impact of social capital on changes in smoking behaviour: a longitudinal cohort study. Eur J Public Health. 2011 Jun;21(3):347-54. doi: 10.1093/eurpub/ckq048. Epub 2010 Jun 21. PMID 20570962
- [Background] Lindstrom M, Isacsson SO, Elmstahl S. Impact of different aspects of social participation and social capital on smoking cessation among daily smokers: a longitudinal study. Tob Control. 2003 Sep;12(3):274-81. doi: 10.1136/tc.12.3.274. PMID 12958387
- [Background] Lindstrom M, Janzon E. Social capital, institutional (vertical) trust and smoking: a study of daily smoking and smoking cessation among ever smokers. Scand J Public Health. 2007;35(5):460-7. doi: 10.1080/14034940701246090. PMID 17852983
- [Background] Centers for Disease Control and Prevention (CDC). Quitting smoking among adults--United States, 2001-2010. MMWR Morb Mortal Wkly Rep. 2011 Nov 11;60(44):1513-9. PMID 22071589
- [Background] Hernandez D, Phillips D. Benefit or burden? Perceptions of energy efficiency efforts among low-income housing residents in New York City. Energy Res Soc Sci. 2015 Jul 1;8:52-59. doi: 10.1016/j.erss.2015.04.010. PMID 27054092
- [Background] Hernandez D, Phillips D, Siegel EL. Exploring the Housing and Household Energy Pathways to Stress: A Mixed Methods Study. Int J Environ Res Public Health. 2016 Sep 14;13(9):916. doi: 10.3390/ijerph13090916. PMID 27649222
- [Background] Gould CF, Chillrud SN, Phillips D, Perzanowski MS, Hernandez D. Soot and the city: Evaluating the impacts of Clean Heat policies on indoor/outdoor air quality in New York City apartments. PLoS One. 2018 Jun 28;13(6):e0199783. doi: 10.1371/journal.pone.0199783. eCollection 2018. PMID 29953529
- [Background] Carrion D, Lee WV, Hernandez D. Residual Inequity: Assessing the Unintended Consequences of New York City's Clean Heat Transition. Int J Environ Res Public Health. 2018 Jan 11;15(1):117. doi: 10.3390/ijerph15010117. PMID 29324717
- [Background] Hernandez D, Swope CB, Azuogu C, Siegel E, Giovenco DP. 'If I pay rent, I'm gonna smoke': Insights on the social contract of smokefree housing policy in affordable housing settings. Health Place. 2019 Mar;56:106-117. doi: 10.1016/j.healthplace.2019.01.007. Epub 2019 Feb 1. PMID 30716667
- [Background] Hernandez D. Affording Housing at the Expense of Health: Exploring the Housing and Neighborhood Strategies of Poor Families. J Fam Issues. 2016 May;37(7):921-946. doi: 10.1177/0192513X14530970. PMID 27057078
- [Background] Hernandez D. "Extra Oomph:" Addressing Housing Disparities through Medical Legal Partnership Interventions. Hous Stud. 2016;31(7):871-890. doi: 10.1080/02673037.2016.1150431. Epub 2016 Apr 13. PMID 27867247
- [Background] Hernandez D. Understanding 'energy insecurity' and why it matters to health. Soc Sci Med. 2016 Oct;167:1-10. doi: 10.1016/j.socscimed.2016.08.029. Epub 2016 Aug 21. PMID 27592003
- [Background] Navas-Acien A, Carkoglu A, Ergor G, Hayran M, Erguder T, Kaplan B, Susan J, Magid H, Pollak J, Cohen JE. Compliance with smoke-free legislation within public buildings: a cross-sectional study in Turkey. Bull World Health Organ. 2016 Feb 1;94(2):92-102. doi: 10.2471/BLT.15.158238. Epub 2015 Nov 23. PMID 26908959
- [Background] Stillman FA, Soong A, Zheng LY, Navas-Acien A. Clear Skies and Grey Areas: Flight Attendants' Secondhand Smoke Exposure and Attitudes toward Smoke-Free Policy 25 Years since Smoking was Banned on Airplanes. Int J Environ Res Public Health. 2015 Jun 4;12(6):6378-87. doi: 10.3390/ijerph120606378. PMID 26053296
- [Background] Apelberg BJ, Hepp LM, Avila-Tang E, Gundel L, Hammond SK, Hovell MF, Hyland A, Klepeis NE, Madsen CC, Navas-Acien A, Repace J, Samet JM, Breysse PN. Environmental monitoring of secondhand smoke exposure. Tob Control. 2013 May;22(3):147-55. doi: 10.1136/tobaccocontrol-2011-050301. Epub 2012 Sep 4. PMID 22949497
- [Background] Jones MR, Wipfli H, Shahrir S, Avila-Tang E, Samet JM, Breysse PN, Navas-Acien A; FAMRI Bar Study Investigators. Secondhand tobacco smoke: an occupational hazard for smoking and non-smoking bar and nightclub employees. Tob Control. 2013 Sep;22(5):308-14. doi: 10.1136/tobaccocontrol-2011-050203. Epub 2012 Jan 24. PMID 22273689
- [Background] Erazo M, Iglesias V, Droppelmann A, Acuna M, Peruga A, Breysse PN, Navas-Acien A. Secondhand tobacco smoke in bars and restaurants in Santiago, Chile: evaluation of partial smoking ban legislation in public places. Tob Control. 2010 Dec;19(6):469-74. doi: 10.1136/tc.2009.035402. Epub 2010 Aug 25. PMID 20798021
- [Background] Stillman F, Navas-Acien A, Ma J, Ma S, Avila-Tang E, Breysse P, Yang G, Samet J. Second-hand tobacco smoke in public places in urban and rural China. Tob Control. 2007 Aug;16(4):229-34. doi: 10.1136/tc.2006.018333. PMID 17652237
- [Background] Navas-Acien A, Peruga A, Breysse P, Zavaleta A, Blanco-Marquizo A, Pitarque R, Acuna M, Jimenez-Reyes K, Colombo VL, Gamarra G, Stillman FA, Samet J. Secondhand tobacco smoke in public places in Latin America, 2002-2003. JAMA. 2004 Jun 9;291(22):2741-5. doi: 10.1001/jama.291.22.2741. PMID 15187056
- [Background] Barnoya J, Navas-Acien A. Protecting the world from secondhand tobacco smoke exposure: where do we stand and where do we go from here? Nicotine Tob Res. 2013 Apr;15(4):789-804. doi: 10.1093/ntr/nts200. Epub 2012 Oct 15. PMID 23072872
- [Background] Moon KA, Rule AM, Magid HS, Ferguson JM, Susan J, Sun Z, Torrey C, Abubaker S, Levshin V, Carkoglu A, Radwan GN, El-Rabbat M, Cohen JE, Strickland P, Breysse PN, Navas-Acien A. Biomarkers of Secondhand Smoke Exposure in Waterpipe Tobacco Venue Employees in Istanbul, Moscow, and Cairo. Nicotine Tob Res. 2018 Mar 6;20(4):482-491. doi: 10.1093/ntr/ntx125. PMID 28582531
- [Background] Jones MR, Navas-Acien A, Yuan J, Breysse PN. Secondhand tobacco smoke concentrations in motor vehicles: a pilot study. Tob Control. 2009 Oct;18(5):399-404. doi: 10.1136/tc.2009.029942. Epub 2009 Aug 25. PMID 19706642
- [Background] Wipfli H, Avila-Tang E, Navas-Acien A, Kim S, Onicescu G, Yuan J, Breysse P, Samet JM; Famri Homes Study Investigators. Secondhand smoke exposure among women and children: evidence from 31 countries. Am J Public Health. 2008 Apr;98(4):672-9. doi: 10.2105/AJPH.2007.126631. Epub 2008 Feb 28. PMID 18309121
- [Background] Apostolou A, Garcia-Esquinas E, Fadrowski JJ, McLain P, Weaver VM, Navas-Acien A. Secondhand tobacco smoke: a source of lead exposure in US children and adolescents. Am J Public Health. 2012 Apr;102(4):714-22. doi: 10.2105/AJPH.2011.300161. Epub 2011 Dec 1. PMID 21852639
- [Background] Soong A, Navas-Acien A, Pang Y, Lopez MJ, Garcia-Esquinas E, Stillman FA. A Cross-Sectional Study of Tobacco Advertising, Promotion, and Sponsorship in Airports across Europe and the United States. Int J Environ Res Public Health. 2016 Sep 28;13(10):959. doi: 10.3390/ijerph13100959. PMID 27690072
- [Background] Branas CC, Cheney RA, MacDonald JM, Tam VW, Jackson TD, Ten Have TR. A difference-in-differences analysis of health, safety, and greening vacant urban space. Am J Epidemiol. 2011 Dec 1;174(11):1296-306. doi: 10.1093/aje/kwr273. Epub 2011 Nov 11. PMID 22079788
- [Background] Kondo MC, Keene D, Hohl BC, MacDonald JM, Branas CC. A Difference-In-Differences Study of the Effects of a New Abandoned Building Remediation Strategy on Safety. PLoS One. 2015 Jul 8;10(7):e0129582. doi: 10.1371/journal.pone.0129582. eCollection 2015. PMID 26153687
- [Background] Giovenco DP, Spillane TE, Merizier JM. Neighborhood Differences in Alternative Tobacco Product Availability and Advertising in New York City: Implications for Health Disparities. Nicotine Tob Res. 2019 Jun 21;21(7):896-902. doi: 10.1093/ntr/nty244. PMID 30452712
- [Background] Giovenco DP, Ackerman C, Hrywna M, Delnevo CD. Changes in the availability and promotion of non-cigarette tobacco products near high schools in New Jersey, USA. Tob Control. 2018 Sep;27(5):578-579. doi: 10.1136/tobaccocontrol-2017-053800. Epub 2017 Aug 10. No abstract available. PMID 28798262
- [Background] Kegler MC, Bundy L, Haardorfer R, Escoffery C, Berg C, Yembra D, Kreuter M, Hovell M, Williams R, Mullen PD, Ribisl K, Burnham D. A minimal intervention to promote smoke-free homes among 2-1-1 callers: a randomized controlled trial. Am J Public Health. 2015 Mar;105(3):530-7. doi: 10.2105/AJPH.2014.302260. Epub 2015 Jan 20. PMID 25602863
- [Background] Sussman JB, Hayward RA. An IV for the RCT: using instrumental variables to adjust for treatment contamination in randomised controlled trials. BMJ. 2010 May 4;340:c2073. doi: 10.1136/bmj.c2073. PMID 20442226
- [Background] Blackstone MM, Wiebe DJ, Mollen CJ, Kalra A, Fein JA. Feasibility of an interactive voice response tool for adolescent assault victims. Acad Emerg Med. 2009 Oct;16(10):956-62. doi: 10.1111/j.1553-2712.2009.00519.x. PMID 19799571
- [Background] Wiebe DJ, Carr BG, Datner EM, Elliott MR, Richmond TS. Feasibility of an automated telephone survey to enable prospective monitoring of subjects whose confidentiality is paramount: a four-week cohort study of partner violence recurrence after Emergency Department discharge. Epidemiol Perspect Innov. 2008 Jan 7;5:1. doi: 10.1186/1742-5573-5-1. PMID 18179709
- [Background] Yancey AK, Ortega AN, Kumanyika SK. Effective recruitment and retention of minority research participants. Annu Rev Public Health. 2006;27:1-28. doi: 10.1146/annurev.publhealth.27.021405.102113. PMID 16533107
- [Background] Brookhart MA, Rassen JA, Schneeweiss S. Instrumental variable methods in comparative safety and effectiveness research. Pharmacoepidemiol Drug Saf. 2010 Jun;19(6):537-54. doi: 10.1002/pds.1908. PMID 20354968
- [Derived] Hernandez D, Khan F, Albert D, Giovenco D, Branas C, Valeri L, Navas-Acien A. A randomized control trial to support smoke-free policy compliance in public housing. Trials. 2023 Aug 22;24(1):551. doi: 10.1186/s13063-023-07339-4. PMID 37608390
- [Derived] Hernandez D, Khan FY, Albert D, Giovenco D, Branas C, Valeri L, Navas-Acien A. A Randomized Control Trial to support smoke-free policy compliance in public housing. Res Sq [Preprint]. 2023 Apr 20:rs.3.rs-2701542. doi: 10.21203/rs.3.rs-2701542/v1. PMID 37131643
- See also: Schoenmarklin S, Consortium TCL. Secondhand smoke seepage into multi-unit affordable housing. St Paul (MN): Tobacco Control Legal Consortium. 2010. — https://publichealthlawcenter.org/sites/default/files/resources/tclc-syn-secondhand-2010.pdf
- See also: U.S. Department of Housing and Urban Development. Instituting Smoke-Free Public Housing. Federal Register; 2016. — https://www.govinfo.gov/content/pkg/FR-2016-12-05/pdf/2016-28986.pdf
- See also: Americans for Nonsmokers' Rights. Smokefree Lists, Maps, and Data. 2017; http://www.no- smoke.org/goingsmokefree.php?id=519, July 1, 2017. — https://no-smoke.org/materials-services/lists-maps/
- See also: American Lung Association. Smoke-free Policies in Multi-Unit Housing - Steps for Success. 2016; http://www.lung.org/our-initiatives/tobacco/smokefree-environments/multi-unit-housing/. Accessed August 4, 2016. — https://www.lung.org/policy-advocacy/tobacco/smokefree-environments/multi-unit-housing
- See also: U.S. Environmental Protection Agency. Secondhand Tobacco Smoke and Smoke-free Homes | Indoor Air Quality (IAQ). 2016; https://www.epa.gov/indoor-air-quality-iaq/secondhand-tobacco-smoke-and- smoke-free-homes. Accessed August 28, 2017. — https://www.epa.gov/indoor-air-quality-iaq/secondhand-smoke-and-smoke-free-homes
- See also: Centers for Disease Control and Prevention. CDC Fact Sheet: Tobacco Industry Marketing. 2016; https://www.cdc.gov/tobacco/data_statistics/fact_sheets/tobacco_industry/marketing/index.htm. Accessed September 30, 2017. — https://www.cdc.gov/tobacco/data_statistics/fact_sheets/tobacco_industry/marketing/index.htm
- See also: Dannenberg AL, Frumkin H, Jackson RJ. Making Healthy Places: Designing and Building for Health, Well-Being, and Sustainability. Berkeley Planning Journal. 2012;25. — https://www.ftc.gov/reports/federal-trade-commission-cigarette-report-2014-federal-trade-commission-smokeless-tobacco
- See also: Greatest engineering achievements of the 20th century. 2003; www.greatachievements.org. Accessed August 28, 2017. — http://www.greatachievements.org
- See also: Leonard TC. Richard H. Thaler, Cass R. Sunstein, Nudge: Improving decisions about health, wealth, and happiness. Constitutional Political Economy. 2008;19(4):356-360. — https://www.google.com/url?sa=t&rct=j&q=&esrc=s&source=web&cd=&ved=2ahUKEwjZkK68mvDxAhUpGFkFHYQgCaoQFjABegQIARAD&url=https%3A%2F%2Fwww.researchgate.net%2Ffile.PostFileLoader.html%3Fid%3D53abe564cf57d7df1e8b45f4%26assetKey%3DAS%253A273548994646025%25401442230571326&usg=AOvVaw0OVZrtfncCZFESGbBqixH4
- See also: U.S. National Cancer Institute. A Socioecological Approach to Addressing Tobacco Related Health Disparities. National Cancer Institute Tobacco Control Monograph 22. NIH Publication No. 17-CA- 8035A. Bethesda, MD: U.S. Department of Health and Human Se — https://cancercontrol.cancer.gov/brp/tcrb/monographs/monograph-22
- See also: Ajzen I. From intentions to actions: A theory of planned behavior. Action control: Springer; 1985. — https://link.springer.com/chapter/10.1007/978-3-642-69746-3_2